CLINICAL TRIAL: NCT04342000
Title: The Effect of Movement Education on Jumping/Landing Quality in High School Athletes: A Randomized Controlled Trial
Brief Title: The Effect of Movement Education on Jumping/Landing Quality in High School Athletes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was updated and is now under IRB #2023-0499
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-1095
Record Dates: First submitted 2020-03-24; First posted 2020-04-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-08

CONDITIONS: ACL Injury
Keywords: movement; education; injury; prevention
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Movement Education Workshop
  Interventions: Other: Movement education workshop
- Control Group (Sham Comparator): Sham Education Workshop
  Interventions: Other: Sham Education Workshop

INTERVENTIONS:
Other: Movement education workshop — 30 minutes total:
  * 10 minutes sedentary activity (LE injury risk factor and anatomy instruction)
  * 10 minutes moderate activity (guided discovery of body segment alignment and stability with squat, lunge, plank, jump, and hop technique assessment and corrective feedback)
  * 10 minutes vigorous activity (practical application of body segment alignment and stability including hopping, jumping, and running activities with technique assessment and corrective feedback)
  For the month following the athlete workshop, prior to the final assessment, subjects will receive periodic text message instructions. These messages will include key facts and takeaways from the workshop, and reminders about correct form.
  Arms: Intervention Group
Other: Sham Education Workshop — 30 minutes total:
  * 10 minute sedentary activity (sleep, nutrition, and hydration instruction)
  * 10 minutes moderate activity (performance of squat, lunge, plank, jump, and hop activities - no technique assessment or corrective feedback)
  * 10 minutes vigorous activity (hopping, jumping, and running activities - no technique assessment and corrective feedback)
  Arms: Control Group

SUMMARY:
While much evidence exists to support the association between physical training and improved motor skill performance, there is little evidence that supports the association between movement education and improved motor skill performance. In short, the investigators would like to study the effect of movement education (as provided by the Sports Safety athlete education program) on immediate and sustained changes in motor skill performance (jumping and landing technique) using the Dynamic Athletic Research Institute (DARI) motion capture system.

This study will evaluate the change in motor performance for high school athletes who did and did not attend the Sport Safety athlete Education Program.

DETAILED DESCRIPTION:
Successful models of injury prevention in occupational health settings focus largely on motor skill education for employees. Sports-related injury prevention programs lack this critical component. This research question is being asked to help inform the development of a comprehensive implementation strategy for a high school sports injury prevention program.

The Hospital for Special Surgery (HSS) Sports Safety ACL Program is a unique, public health approach to ACL injury risk management. The program offers pioneering education to those directly responsible for the safety of young athletes. The program offers diverse educational opportunities and innovative risk management resources directly to coaches, parents, administrators, and young athletes. The program has already held over 200 live workshops, teaching coaches, parents and young athletes how to identify injury risk factors and how the relationship between movement quality and sports performance impacts injury rates. Though several research studies have been conducted with the HSS Sport Safety Program, this study is the first to evaluate the association between athlete motor learning and movement quality.

Currently anterior cruciate ligament (ACL) injury prevention programs focus on clinicians and coaches leading a series of neuromuscular training exercises repeatedly throughout a sports season to improve athlete strength, balance, flexibility, and agility. While this has shown been shown to be effective in controlled research settings, there have been many problems with implementation, including low compliance. Hartigan et al recently conducted a study showing that athletes had improved jumping and landing technique after viewing video feedback. This is evidence that movement education/feedback has the ability to affect motor skills. Demonstrating an association between motor skill education and improved movement quality would allow the responsibility of ACL injury prevention to be more readily shared by both sports medicine clinicians and athletes.

This evidence would provide support for the public health approach to ACL injury risk management on which the HSS Sport Safety Program was based. In addition, providing solid evidence of the program's success will make the program more marketable to schools, clubs, and other sports groups nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18
* Participates in a high-risk sport for ACL injury (e.g. basketball, soccer, lacrosse)

Exclusion Criteria:

* Current injuries that would interfere with ability to perform vertical, box, broad jumps
* History of knee injuries or surgeries

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Dynamic Valgus Degrees | Change from baseline to immediately following intervention (average of 30 minutes after baseline),1 month after baseline
  dynamic valgus degrees in vertical jump as measured by DARI
Dynamic Valgus Depth | Change from baseline to immediately following intervention (average of 30 minutes after baseline),1 month after baseline
  dynamic valgus depth in cm in vertical jump as measured by DARI

SECONDARY OUTCOMES:
Athlete education outcomes | Change from baseline to immediately following intervention (average of 30 minutes after baseline),1 month after baseline
  as measured by pre- and post-education surveys

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Marx, MD, Principal Investigator — Hospital for Special Surgery, New York

IPD SHARING:
Plan to Share IPD: No